CLINICAL TRIAL: NCT03860896
Title: A Phase 1b, Randomized, Double-blind, Placebo-controlled, Multi-center Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of GB004 in Adult Subjects With Active Ulcerative Colitis
Brief Title: GB004 in Adult Subjects With Active Ulcerative Colitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GB004, Inc., a wholly owned subsidiary of Gossamer Bio, Inc. (Industry)
Responsible Party: Sponsor
Organization: Gossamer Bio Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GB004-1101
Record Dates: First submitted 2019-02-14; First posted 2019-03-04 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Ulcerative Colitis
Keywords: Inflammatory Bowel Disease; Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GB004 (Experimental): GB004 for oral administration daily
  Interventions: Drug: GB004
- Placebo (Placebo Comparator): Placebo for oral administration daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GB004 — GB0004 high dose
  Arms: GB004
Drug: Placebo — Placebo
  Arms: Placebo
Drug: GB004 — GB004 low dose
  Arms: GB004

SUMMARY:
This is a Phase 1b, randomized, double-blind-, placebo-controlled, multi-center study to evaluate the safety, tolerability, and PK of GB004 in adult subjects with active ulcerative colitis. Target engagement and effect of GB004 on pharmacodynamic biomarkers will be assessed.

DETAILED DESCRIPTION:
The safety, tolerability, pharmacokinetics, and pharmacodynamics of GB004 will be explored in a Phase 1b randomized controlled trial in adults subjects with active ulcerative colitis (UC). Subjects will be evaluated based on incidence of AEs, laboratory parameters, GB004 serum and colonic tissue concentrations, and changes in the signs and symptoms of UC.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-74, receiving therapy for active ulcerative colitis confirmed by Mayo Score assessment, and evidence of colonic inflammation.

Exclusion Criteria:

* Evidence of Crohn's disease, indeterminate colitis, or presence of bacterial or parasitic infection.
* Patients receiving biologic agents and experimental agents are excluded.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-04-24 (Actual); Primary Completion 2019-12-17 (Actual); Study Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | 56 Days
  To evaluate the safety and tolerability of GB004 for 56 days in terms of incidence of treatment emergent adverse events reported.

SECONDARY OUTCOMES:
Pharmacokinetics: Time to Reach Maximum Concentration (Tmax) of GB004 | Day 1 to Day 28
Pharmacokinetics: Maximum Concentration (Cmax) of GB004 | Day 1 to Day 28
Pharmacokinetics: Area Under the Concentration Curve (AUC) of GB004 | Day 1 to Day 28

CONTACTS AND LOCATIONS:
Locations (3):
- Delta Research Partners, Monroe, Louisiana, United States
- Arensia Exploratory Medicine, Tbilisi, Georgia
- PMSI Republican Clinical Hospital "Timofei Mosneaga", Chisinau, Moldova

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Danese S, Levesque BG, Feagan BG, Jucov A, Bhandari BR, Pai RK, Taylor Meadows K, Kirby BJ, Bruey JM, Olson A, Osterhout R, Van Biene C, Ford J, Aranda R, Raghupathi K, Sandborn WJ. Randomised clinical trial: a phase 1b study of GB004, an oral HIF-1alpha stabiliser, for treatment of ulcerative colitis. Aliment Pharmacol Ther. 2022 Feb;55(4):401-411. doi: 10.1111/apt.16753. Epub 2022 Jan 10. PMID 35014040